CLINICAL TRIAL: NCT00002186
Title: Double-Blind Placebo-Controlled Study Comparing the Combination of 15% SP-303 Gel With Acyclovir Versus Acyclovir Alone for the Treatment of Recurrent Herpes Simplex Virus (HSV) Infections in Subjects With Acquired Immunodeficiency Syndrome (AIDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaman Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 270A; 96-867-DE
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-02

CONDITIONS: Herpes Simplex; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Herpes Simplex; Drug Therapy, Combination; Acyclovir; Antiviral Agents; Gels; SP 303
MeSH Terms: conditions — Herpes Simplex; HIV Infections; AIDS-Related Opportunistic Infections | interventions — crofelemer; Acyclovir

INTERVENTIONS:
Drug: Crofelemer
Drug: Acyclovir

SUMMARY:
To evaluate the safety of topically applied SP-303 gel and to compare the efficacy of SP-303 gel in combination with acyclovir, relative to acyclovir alone, for the treatment of recurrent Herpes Simplex Virus (HSV) 1 and 2 infections, affecting the genital, perianal and neighboring areas, in patients with AIDS.

DETAILED DESCRIPTION:
This trial is a double-blind, multicenter, placebo-controlled clinical trial. Participants are randomized to topical 15% SP-303 gel and oral acyclovir or to matching topical placebo gel and oral acyclovir. At presentation, patients are stratified by total lesion area within each treatment group. SP-303 or matching placebo is topically applied three times a day until all lesions are reepithelialized or for 14 days, whichever occurs earlier. Acyclovir is administered by mouth each day, three times a day, until all lesions are reepithelialized or for 14 days, whichever occurs earlier. Patients are evaluated for lesion healing and adverse events 3 times per week during the treatment period. The primary efficacy endpoint will be complete lesion healing and the primary analysis will be time to complete healing.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* AIDS, according to the CDC criteria.
* Documented recurrent (at least 1 prior episode) perineal (genital, perianal and neighboring areas) mucocutaneous herpes simplex virus (HSV) types 1 or 2 infection in the active phase.
* Duration of current episode of recurrent HSV lesions of 3 days or less.
* Ability to read and write, must be intellectually competent, and able to understand the purposes and risks of the study.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Active internal anal or rectal herpes.
* Inability to comply with protocol.
* Impaired renal function.

Patients with the following prior conditions are excluded:

* Prior episode of recurrent genital herpes infection with documented clinical failure of acyclovir as a treatment regimen.
* Uncompensated hepatic, cardiac, or renal failure within 1 month of the study.
* History of hypersensitivity to acyclovir.
* Previous enrollment in this study.

  1. Treatment with another medication (topical, oral, or intravenous) with known anti-HSV activity within the past 5 days.
* Systemic immunomodulatory therapy within 30 days prior to study.
* Previous treatment with SP-303.

Required:

Unchanged antiretroviral therapy for the 2 weeks prior to study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400

CONTACTS AND LOCATIONS:
Locations (34):
- United States (32):
  - Sorra Research Ctr Inc / Med Forum, Birmingham, Alabama
  - Hill Top Research Ltd, Scottsdale, Arizona
  - Arizona Clinical Research Ctr Inc, Tucson, Arizona
  - Dermatology SVC - VAMC, Long Beach, California
  - King - Drew Med Ctr / Dept of Dermatology, Los Angeles, California
  - Summit Med Ctr / Adult Immunology Clinic, Oakland, California
  - ViRx Inc, Palm Springs, California
  - ViRx Inc, San Francisco, California
  - Conant Med Ctr, San Francisco, California
  - Olive View Med Ctr, Sylmar, California
  - Novum Inc, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Gary Richmond MD, Fort Lauderdale, Florida
  - Dr Robert Schwartz, Fort Myers, Florida
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - Veterans Affairs Med Ctr of North Chicago, Chicago, Illinois
  - Johns Hopkins Univ / Division of Infectious Disease, Baltimore, Maryland
  - Saint Agnes Healthcare / Dept of Surgery, Baltimore, Maryland
  - Massachusetts Gen Hosp - Warren 505, Boston, Massachusetts
  - Medicine / Infectious Diseases, Minneapolis, Minnesota
  - AIDS Ctr / Saint Vincents Hosp and Med Ctr, New York, New York
  - New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Paddington Testing Co Inc, Philadelphia, Pennsylvania
  - Austin Infectious Disease Consultants, Austin, Texas
  - N Texas Ctr for AIDS & Clin Rsch, Dallas, Texas
  - Division of Infectious Diseases / Univ of Texas - Houston, Houston, Texas
  - Dr Robert Holman, Arlington, Virginia
  - Novum Inc, Seattle, Washington
  - Univ of Washington Virology Research Clinic, Seattle, Washington
- Puerto Rico (2):
  - Hosp Regional de Ponce - Area Vieja, Ponce
  - San Juan AIDS Program, Santurce